CLINICAL TRIAL: NCT05980299
Title: Testing the Feasibility of the Individualized Positive Psychosocial Intervention (IPPI)
Acronym: IPPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Collaborators: United Church Homes (Unknown); Penn State University (Other); Virginia Polytechnic Institute and State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FY22_Pilot5_Abbott; U54AG063546 (NIH); 403853 (Other: Miami University Index)
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Depression; Behavior
Keywords: dementia; depressive symptoms; psychosocial intervention; feasibility; emotion
MeSH Terms: conditions — Dementia; Depression; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): The experimental arm involves a brief positive interaction around a preferred activity or personal care routine.
  Interventions: Behavioral: Individualized Positive Psychosocial Interaction

INTERVENTIONS:
Behavioral: Individualized Positive Psychosocial Interaction — The intervention involves a brief positive interaction around a preferred activity or personal care routine.
  Other Names: Individualized Positive Psychosocial Intervention

SUMMARY:
The goal of this clinical trial is to test the feasibility of the Individualized Positive Psychosocial Interaction (IPPI) with 108 nursing home residents living with dementia and distress or depressive symptoms. The main questions it aims to answer are: •is it feasible to deliver the IPPI and track impact through data collected in the electronic medical records. Care partners will engage eligible residents in 2 brief preference-based IPPIs per week over the course of 6 months.

DETAILED DESCRIPTION:
Specific Aims. Psychological and behavioral symptoms of distress (BPSD) expressed by people living with dementia (PLWD) are challenging to respond to in nursing home (NH) care. Experienced by 78% of PLWD, BPSD can include wandering, persistent vocalizations, and resistance or refusal of care.1 In addition, 30% of NH residents experience depressive symptoms2 and among those with depressive symptoms, 47% also have dementia.3 Together, these conditions will be referred to as distress throughout this proposal. Without appropriate guidance or training, care partners (e.g., Certified Nursing Assistants) struggle to prevent or positively remediate distress experienced by PLWD. The Individualized Positive Psychosocial Intervention (IPPI) is an evidence-based program designed to support care partners in engaging PLWD with brief (i.e.,10 minute) one-to-one preference-based activities. IPPI is designed to enhance well-being and reduce negative emotional and behavioral responses using non-pharmacological approaches that align care with residents' preferences recorded in Section F of the MDS (e.g., choose what clothes to wear). Specifically, in our IPPI randomized controlled trial (RCT) effectiveness trial,4 NH residents receiving the IPPI program delivered by care partners experienced more pleasure, alertness, engagement, and positive verbal behavior compared with the usual care group.

Our goal with this proposal is to partner with United Church Homes (UCH), a 106-year-old nonprofit national senior living provider to conduct a full implementation feasibility pilot of the IPPI program with long-stay residents in 9 of their NHs. Our objective is to conduct a pilot study to evaluate 1) the ability of staff to identify residents who are optimal for the IPPI, 2) implementation of IPPI, and 3) the impact on pragmatic clinical outcome measures (BPSD and depressive symptoms). Staff champions will be identified by the stakeholder team in each NH (e.g., Director of Nursing, Activity Professional) and trained to identify residents optimal for the IPPI (i.e., experiencing cognitive impairment (Minimum Data Set (MDS) Brief Inventory for Mental Status (BIMS) score 0-12) as well as documentation (MDS Section E or D) of distress within the past 3-months. Distress is indicated by a 1 or higher on any of the 5 behavior items from MDS Section E (i.e., physical, verbal, other behavior, rejection of care, wandering) and/or a score of 1 or higher on one of 5 MDS section D items (i.e., anhedonia, sad mood, poor self-esteem, poor appetite, restlessness).

Care partners of identified residents will be invited to be trained to deliver IPPI. The investigators anticipate that each NH will initiate engagement with 4-5 residents per month for each of 3 consecutive months (12-15 residents per NH) in addition to 3-4 care partners who will deliver the IPPI. Resident initiation in the program will occur on a rolling basis (i.e., initiating intervention activities for a given resident when he/she is due for a routine quarterly care plan review). Each selected resident will then receive 2 IPPI sessions per week for 6 months. The project seeks to achieve the following specific aims:

Aim 1. To conduct a pilot embedded Pragmatic Clinical Trial (ePCT) to evaluate and establish the feasibility of implementing the IPPI program in 9 NHs among 108-135 residents. Quantitative implementation endpoints indicating success include (a) that staff in each community will be able to identify and engage 12-15 residents experiencing both dementia (e.g., BIMS 0-12) and distress (either BPSD or depressive symptoms) within the past 2 weeks, measured by a count of participants; (b) that all the implementation team members (champions and care partners) can complete the online training within the first two months of initiating implementation, as indicated by the learning management system; (c) that the implementation team will be able to (i) review existing data from Section F of the MDS for all selected residents; (ii) identify a match between a resident's important preferences and 1-2 IPPI protocols; (iii) identify a targeted expression of distress as measured by documentation in the electronic medical record; and (d) that staff can conduct at least 2 ten-minute sessions per week, per targeted resident with fidelity over the course of 6 months as measured in the electronic medial record (EMR). Qualitative data to evaluate implementation will be ascertained from semi-structured interviews with implementation team members in each community to assess acceptability, feasibility, and appropriateness as well as facilitators and barriers to fidelity of the IPPI sessions.

Aim 2. To establish the feasibility of tracking intervention impact on a primary clinical outcome of a targeted behavior (identified by staff) through the MDS Section E (E0200A, B or C; or E0800) or MDS Section D (Patient Health Questionnaire (PHQ-9) items of anhedonia, sad mood, poor self-esteem, poor appetite, or restlessness). The primary outcome measure will consist of a single variable indicating improvement, no change, or worsening of a staff-targeted behavior of distress of each resident receiving the intervention, tracked pre- and post-IPPI intervention using routinely collected data in the EMR. Secondary staff outcomes will include knowledge of emotion-focused communication and staff reported self-efficacy in applying the communication skills.

IMPACT: The IPPI program teaches care partners strategies to better identify and manage their own feelings and those of PLWD through our emotion-focused communication course. In addition, the program provides highly structured and feasible protocols to guide short but impactful interactions with PLWD designed to prevent and remediate distress (i.e., BPSD and symptoms of depression). Findings from this pilot study will guide the implementation, approach, and power needed for a full-scale Stage IV effectiveness ePCT study.

ELIGIBILITY:
Inclusion Criteria:

Eligibility for Individualized Positive Psychosocial Interaction (IPPI)

1. Be a long-term resident in a nursing home
2. Have a score of 0-12 on the Brief Inventory for Mental Status (BIMS)
3. Either (could be both) on their most recent Minimum Data Set (MDS) 3.0 assessment A score of 1 or higher on any of the 5 behavior items from MDS Section E (i.e., physical, verbal, other behavior, rejection of care, wandering) A score of 1 or higher on one of 5 MDS section D items (i.e., anhedonia, sad mood, poor self-esteem, poor appetite, restlessness)

Exclusion Criteria: Nursing home residents who are expected to live in the community for less than 6 months.

-

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Abbott, PhD, Principal Investigator — Miami University
Locations (7):
- United States (7):
  - The Trinity Community at Beavercreek, Beavercreek, Ohio
  - The Chapel Hill Community, Canal Fulton, Ohio
  - The Trinity Community at Fairborn, Fairborn, Ohio
  - The Four Winds Community, Jackson, Ohio
  - The Harmar Place Community, Marietta, Ohio
  - SEM Haven, Milford, Ohio
  - The Parkvue Community, Sandusky, Ohio

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPT) available.

REFERENCES:
- [Background] Van Haitsma KS, Curyto K, Abbott KM, Towsley GL, Spector A, Kleban M. A randomized controlled trial for an individualized positive psychosocial intervention for the affective and behavioral symptoms of dementia in nursing home residents. J Gerontol B Psychol Sci Soc Sci. 2015 Jan;70(1):35-45. doi: 10.1093/geronb/gbt102. Epub 2013 Dec 4. PMID 24304555
- [Result] Abbott KM, Heid AR, Noble M, Kotterman A, Unroe K, Van Haitsma K. An Embedded Pragmatic Clinical Trial of the Individualized Positive Psychosocial Interaction (IPPI) Program. J Am Med Dir Assoc. 2025 Aug;26(8):105700. doi: 10.1016/j.jamda.2025.105700. Epub 2025 Jun 12. PMID 40460889
- See also: IPPI program — https://www.preferencebasedliving.com/ippi/individualized-positive-psychosocial-intervention-protocol-ippi/

RESULTS

PARTICIPANT FLOW:
Groups:
- Staff Care Partners: Staff delivering the IPPIs
Period: Overall Study
Arm/Group | experimental | Staff Care Partners
Started | 130 | 70
Completed | 93 | 60
Not Completed | 37 | 10
Not completed — Death | 28 | 0
Not completed — Discharged from Nursing Home | 9 | 0
Not completed — Lost to Follow-up | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Staff Care partner: staff care partners delivering the IPPI
- Total: Total of all reporting groups
Arm/Group | experimental | Staff Care partner | Total
Number analyzed (Participants) | 130 | 70 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Results for each Arm/Group are presented in separate Rows
  years
    Resident: number analyzed (Participants) | 130 | 0 | 130
    Resident | 84.44 (8.21) |  | 84.44 (8.21)
    Staff Care Partner: number analyzed (Participants) | 0 | 70 | 70
    Staff Care Partner |  | 40.35 (13.94) | 40.35 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 63 | 159
  Male | 34 | 7 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 117 | 64 | 181
  Unknown or Not Reported | 12 | 1 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 4 | 4
  White | 117 | 61 | 178
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 11 | 2 | 13
Marital Status [Count of Participants; unit: Participants] — Population: We did not ask staff care partners about their marital status
  Participants
    Never Married | 9 | 0 | 9
    Married | 31 | 0 | 31
    Widowed | 70 | 0 | 70
    Divorced | 19 | 0 | 19
    Missing | 1 | 70 | 71
Length of Stay [Mean (Standard Deviation); unit: Months] — Number of months residing in nursing home Population: This variable is not applicable for staff care partners
  Months
    number analyzed (Participants) | 130 | 0 | 130
    (all) | 16.79 (22.18) |  | 16.79 (22.18)
Cognition [Mean (Standard Deviation); unit: units on a scale] — Brief Interview for Mental Status (BIMS) is a scale that ranges from 0-15 with higher values indicating more cognitive capacity and 0-12 indicating cognitive impairment. For our sample, the range was 0-12. Population: Variable not applicable for Staff Care Partners
  units on a scale
    number analyzed (Participants) | 130 | 0 | 130
    (all) | 4.68 (3.64) |  | 4.68 (3.64)

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Behavioral Symptoms Directed Toward Others
Description: The investigators are using a person-centered outcome measure. If the participant has an indicate of 1 or more on any of the following items that indicate distress at baseline: Minimum Data Set (MDS) Section E or MDS Section D (Patient Health Questionnaire (PHQ-9). The investigators looked at the same variable 6 months later to see if the symptom remained stable, improved, or worsened.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 18
Participants
  Symptoms stayed stable | 4
  symptoms improved | 13
  symptoms worsened | 1

2. Primary Outcome: Change in Verbal Behavior Symptoms Directed Towards Others
Description: as for outcome 1
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 20
Participants
  Symptoms stayed stable | 5
  symptoms improved | 12
  symptoms worsened | 3

3. Primary Outcome: Change in Other Behavioral Symptoms Not Directed Towards Others
Description: as for outcome 1
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 18
Participants
  Symptoms stayed stable | 0
  symptoms improved | 18
  symptoms worsened | 0

4. Primary Outcome: Change in Rejection of Care
Description: as for outcome 1
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 13
Participants
  Symptoms stayed stable | 5
  symptoms improved | 8
  symptoms worsened | 0

5. Primary Outcome: Change in Wandering
Description: as for outcome 1
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 12
Participants
  Symptoms stayed stable | 3
  symptoms improved | 8
  symptoms worsened | 1

6. Primary Outcome: Change in Little Interest or Pleasure in Doing Things
Description: The investigators are using a person-centered outcome measure. If the participant has an indicate of 1 or more on any of the following items that indicate distress: Minimum Data Set (MDS) Section E (E0200A, B or C; or E0800) or MDS Section D (Patient Health Questionnaire (PHQ-9)
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 18
Participants
  Symptoms stayed stable | 3
  symptoms improved | 15
  symptoms worsened | 0

7. Primary Outcome: Change in Feeling Down, Depressed or Hopeless
Description: as for outcome 1
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | experimental
Number analyzed (Participants) | 23
Participants
  Symptoms stayed stable | 2
  symptoms improved | 20
  symptoms worsened | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definitions do not differ
Groups:
- Staff care partners: Staff completing an emotion-focused communication training and facilitating IPPIs with residents
  Staff Care Partners were not assessed for All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events
Arm/Group | experimental | Staff care partners
All-Cause Mortality (participants affected / at risk) | 28/130 | 0/0
Serious Adverse Events (participants affected / at risk) | 28/130 | 0/0
Other Adverse Events (participants affected / at risk) | 0/130 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | experimental (N=130) | Staff care partners (N=0)
Advanced Dementia (General disorders) | 28 (28) | 0 (0) — 28 individuals passed away due to advanced dementia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT05980299/Prot_SAP_000.pdf